CLINICAL TRIAL: NCT00128206
Title: Clinical Trial of Short Course Rifampin Versus INH for LTBI in Jail
Brief Title: Treatment of Latent TB Infection for Jailed Persons
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-135; U01AI051315 (NIH)
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Tuberculosis
Keywords: LTBI, tuberculosis, rifampin, isoniazid, prisoners
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): isoniazid (INH) (900 mg orally) given twice weekly for 9 months
  Interventions: Drug: Isoniazid
- A (Active Comparator): rifampin (600 mg orally) given daily for 4 months
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Isoniazid — Isoniazid 900 mg twice weekly
  Arms: B
Drug: Rifampin — Rifampin 600mg once per day
  Arms: A

SUMMARY:
The purpose of this study is to determine whether an alternative drug, (rifampin) given daily, is better at treating tuberculosis (TB) and more tolerable than the usual drug treatment, isoniazid (INH). Study participants will include 972, TB infected, San Francisco Jail inmates, aged 18 or older. One group of volunteers will take INH two times a week for 9 months, and the other group will take rifampin daily for 4 months. Medication will be administered in jail and at the San Francisco TB Clinic if the volunteer is released from jail prior to completing the study. Participants will be seen daily for 4 months (rifampin group), and 2 times a week for 9 months (INH group) for directly observed therapy. Study procedures will include 5 symptom review visits and blood samples for lab testing. Follow-up will continue for each subject for five years after enrollment into the study.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate the effect of two accepted regimens for treating latent tuberculosis infection (LTBI) in jail. Tuberculosis (TB) in incarcerated populations continues to be a serious problem, due to the large proportion of persons who are at high risk of both having latent tuberculosis infection (LTBI) and developing active disease. Completion of treatment of LTBI, while an important component of overall TB control efforts, has not been successful in jails. This is primarily because inmates are frequently released before finishing a 6-9 month course of standard therapy, and have low rates of completing therapy in the community. This study proposes to look at toxicity and adherence for this 4-month regimen compared to the nine-month regimen of to isoniazid (INH), and to examine costs, both cost of delivered care and the cost of TB disease prevented, with examination of reasons for completion or noncompletion of therapy. Short-course therapies for LTBI may address this problem but they are more expensive and have not been studied adequately to answer questions about side effects, completion rates, and overall cost. The investigators propose a randomized trial to test the effects of a short course therapy, rifampin (600 mg orally) given daily for 4 months, as compared to (INH) (900 mg orally) given twice weekly for 9 months. Both regimens are listed by the Centers for Disease Control and Prevention (CDC) and the American Thoracic Society as acceptable treatments for persons with LTBI. The study participants will include 972 San Francisco Jail inmates, 18 years and older, enrolled over a 28-month period, for a sample of 486 in each study group. Subjects, followed in jail and after release, will be followed to test three hypotheses: the null hypothesis of a difference in toxicity of rifampin as compared to INH within a 95% confidence interval of (.4-1.87) and no difference by study group in adherence and in cost-effectiveness. A secondary aim is to describe reasons for completion or noncompletion of therapy. Toxicity is defined as complications leading to stopping drug. Adherence is defined as completion of care, or 120 doses taken within 6 months for the rifampin group and 76 doses of INH taken within 12 months for the INH group. Cost effectiveness will be calculated as the total cost of care (nursing, medical, laboratory, as well as facility costs), and measured against costs of TB cases prevented. All treatments will be administered by directly observed therapy (DOT) in jail, and by DOT after release at the San Francisco TB Clinic. Counseling on adherence (going to the TB Clinic if released before completing therapy) and on possible side effects will be given to all study subjects at enrollment and during follow-up clinic visits. All subjects will be routinely evaluated by study personnel every two weeks for the first 6 weeks, and thereafter to detect possible drug toxicity including hepatitis, peripheral neuropathy, arthralgias, rash, memory loss, and other clinical symptoms. All patients will undergo laboratory assessment at regular intervals according to a schedule which compares study group participation and the usual care in the jail. All blood test results, and new symptoms or changes in symptoms found at follow-up, will be added to the jail medical record. A final interview will be done with subjects at the time that they have completed or not completed this course of therapy for LTBI, to determine reasons (barriers and enablers). Follow-up will continue for each subject for five years after enrollment into the study, to measure study endpoint (completion of care, taken off drugs for toxicity or loss to follow-up) and to measure subsequent treatment for LTBI or development of active TB by record review.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for this study will be San Francisco Jail inmates, age 18 or older (the jail does not house juveniles) having evidence of M. tuberculosis infection by positive tuberculin skin test (a documented reactive tuberculin skin test to 0.1 mL containing 5 Tuberculin Units) who meet current national criteria for therapy for tuberculosis infection and can provide informed consent.

Exclusion Criteria:

* Ineligible for either therapy regimen for any of the following reasons:

  1. history of treatment-limiting reaction to isoniazid or rifamycins;
  2. pregnancy or breast feeding;
  3. active tuberculosis;
  4. an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the upper limit of normal;
  5. bilirubin >2 times the upper limit of normal;
  6. platelets <150 K/mm3;
  7. taking protease inhibitors or nonnucleoside reverse transcriptase inhibitors (NNRTIs);
* Unable to communicate in English or Spanish;
* Unable or unwilling to provide informed consent;
* Not in the routine level of jail security for any reason (housed in "special security" areas);
* Any condition that, in the best judgment of the investigator, would pose a risk to the subject during the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2004-11; Primary Completion 2008-10 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary C White, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] White MC, Tulsky JP, Lee JR, Chen L, Goldenson J, Spetz J, Kawamura LM. Isoniazid vs. rifampin for latent tuberculosis infection in jail inmates: toxicity and adherence. J Correct Health Care. 2012 Apr;18(2):131-42. doi: 10.1177/1078345811435973. Epub 2012 Mar 14. PMID 22419641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inmates in the San Francisco City and County Jail diagnosed with latent tuberculosis infection (LTBI) at jail entry were recruited,consented and enrolled between 11/30/2004 and 9/24/2007.
Pre-assignment Details: Of 416 inmates with LTBI who consented to be enrolled, 52 were not randomized because of abnormal liver function tests (20), they were released before they could be assigned to a group (30), or they subsequently changed their mind and refused participation (2).
Groups:
- Isoniazid: isoniazid (INH) (900 mg orally) given twice weekly for 9 months
- Rifampin: rifampin (600 mg orally) given daily for 4 months
Period: Overall Study
Arm/Group | Isoniazid | Rifampin
Started | 184 | 180
Completed | 47 | 60
Not Completed | 137 | 120
Not completed — Lost to Follow-up | 137 | 118
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isoniazid | Rifampin | Total
Number analyzed (Participants) | 184 | 180 | 364
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 180 | 363
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.34 (9.59) | 31.51 (9.57) | 30.9 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 173 | 166 | 339
Region of Enrollment [Number; unit: participants]
  United States | 184 | 180 | 364

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Laboratory Test or Clinical Judgment Resulting in the Need to Stop Study Medication
Description: Liver function tests were taken at regular intervals and clinical symptoms were reviewed at regular intervals in both study groups. On the basis of these tests and examinations, physicians determined whether the study drug needed to be stopped.
Time Frame: up to one year
Population: The number of participants was determined by power calculations using estimates of toxicity from the literature. The analysis was intention to treat.
Measure: Number; unit: participants
Arm/Group | Isoniazid | Rifampin
Number analyzed (Participants) | 184 | 180
participants | 6 | 3
Statistical Analysis 1: Comparison: Isoniazid vs Rifampin; The null hypothesis was that there would be no difference in toxicity by study group, and a sample of 360 participants (180 in each group)was estimated to have sufficient power to detect a difference; Test type: Superiority or Other; p > .05, Chi-squared; Risk Ratio (RR) = .51, 95% CI [.13 to 2.01]

2. Secondary Outcome: Completion of Therapy
Time Frame: course of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Isoniazid | Rifampin
Number analyzed (Participants) | 184 | 180
Participants | 47 | 60

3. Secondary Outcome: Cost Effectiveness
Time Frame: course of treatment
Population: Cost effectiveness data were not collected.
Arm/Group | Isoniazid | Rifampin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the course of treatment for each participant, until treatment was completed or subject was lost or withdrawn from the study. This was up to 1 year for all participants.
Description: Participants had routine blood tests for liver functions and clinical review for symptoms at regular intervals during receipt of the study medication. While they remained in jail, adverse events also were collected for all sick call visits to jail health personnel.
Arm/Group | Isoniazid | Rifampin
Serious Adverse Events (participants affected / at risk) | 11/184 | 3/180
Other Adverse Events (participants affected / at risk) | 46/184 | 45/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isoniazid (N=184) | Rifampin (N=180)
elevated liver function test (Hepatobiliary disorders) | 8 (8) | 1 (1)
suicidal thoughts (Psychiatric disorders) | 1 (1) | 1 (1)
hospitalization for ankle surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
hospitalization for appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
allergic reaction (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Isoniazid (N=184) | Rifampin (N=180)
gastrointestinal symptoms (Gastrointestinal disorders) | 12 | 10
skin rash (Skin and subcutaneous tissue disorders) | 13 | 16
elevated liver function tests (Hepatobiliary disorders) | 12 | 8
injury (Injury, poisoning and procedural complications) | 9 | 11 — injury from athletic activities or fights or accidents in the jail

LIMITATIONS AND CAVEATS:
Initial enrollment estimates were not met, from lower TB rates, increased deportation rates and fewer Jail personnel for LTBI testing. The complexity of treatment in the jail led to technical problems in the analytic plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes